CLINICAL TRIAL: NCT00000873
Title: A Randomized, Double-Blind, Controlled Study of an Increased Caloric Density Infant Formula and Its Effect on Growth and Nutritional Status in HIV-Infected Infants
Brief Title: A Study on the Effect of High-Calorie Infant Formula on Growth and Nutrition in HIV-Infected Infants
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: National Institute of Allergy and Infectious Diseases (NIAID) (NIH)
Collaborators: Eunice Kennedy Shriver National Institute of Child Health and Human Development (NICHD) (NIH)
Responsible Party: Sponsor
Model: Parallel | Purpose: Treatment
Other Study IDs: ACTG 247; PACTG 247; ACTG 844 Substudy; 11224 (Registry Identifier: DAIDS ES)
Record Dates: First submitted 1999-11-02; First posted 2001-08-31 (Estimated); Last update posted 2013-10-07 (Estimated); Status verified 2013-10

CONDITIONS: HIV Infections
Keywords: Nutritional Status; HIV Seronegativity; Infant Food
MeSH Terms: conditions — HIV Infections | interventions — Infant Formula

INTERVENTIONS:
Drug: Infant Formula

SUMMARY:
This study examines the effects of an infant formula containing increased calories, as compared to commercial formulas, when given during the first 6 months of life. It will examine effects on growth, disease progress, immune system, and quality of life of infected infants.

HIV disease in infants often leads to nutritional deficiencies. Providing increased nutrition early in their lives may help the quality of life of children who contract HIV from their mothers.

DETAILED DESCRIPTION:
In order to meet the optimal nutritional needs of HIV-infected infants, it is critical that nutritional intervention begin early. Early nutritional intervention may help reduce the susceptibility to or severity of primary HIV and/or opportunistic infections and add to the quality of life for children perinatally infected with HIV.

[AS PER AMENDMENT 08/29/01: This study population will consist of infants from domestic sites and international sites.] In this double-blind, controlled study perinatally HIV-exposed infants less than 15 days old [AS PER AMENDMENT 08/29/01: "less than 15 days old" has been replaced with: less than 17 days old] at time of study entry are randomized to 1 of 2 arms to receive either concentrated formula or standard formula for 8 weeks after being stratified by gestational age: less than 37 versus greater than 37 completed weeks. At the 8-week visit using a previously determined 8:1 random allocation, 89% of singleton infants [AS PER AMENDMENT 08/29/01: from international sites] with negative HIV-specific tests are discontinued from study treatment and further follow-up. The other 11 percent of these singleton infants with negative HIV-specific tests continue study treatment with open-label standard formula until Week 28 (control group). Singleton infants with positive HIV-specific tests continue on the blinded portion of the study and receive formula as initially assigned until Week 28. For a given multiple birth, if any of the infants at the 8-week study visit are determined to be infected, all the infants from that birth continue their initial blinded treatment assignment until Week 28; if none of the infants are determined to be infected at this time, all the infants from that birth continue study treatment with open-label standard formula until Week 28. All infants assigned to receive study treatment through Week 28 continue study follow-up until 12 months of age. A subset of patients at sites with appropriate resources will participate in a substudy in which measurements of triceps and thigh skinfold thickness and circumference and thigh density DEXA scans are evaluated.

ELIGIBILITY:
Inclusion Criteria

Children may be eligible for this study if they:

* Are 1 to 17 days old. (This study has been changed. Originally, infants 1 to 15 days old were eligible for this study.)
* Weigh 4 or more pounds.
* Were born to an HIV-positive mother.
* Have a caregiver willing to measure and keep records of infant's food intake.

Exclusion Criteria

Children will not be eligible for this study if they:

* Are breast-fed.
* Have certain disorders, including the inability to feed by mouth, or a life-threatening condition.
* Take medication which affects growth.

Ages: 1 Day to 17 Days | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 2400
Dates: Study Completion 2005-09 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Harland S Winter, Study Chair; James Oleske, Study Chair; Ross McKinney, Study Chair
Locations (72):
- United States (62):
  - Univ of Alabama at Birmingham - Pediatric, Birmingham, Alabama
  - Univ of South Alabama, Mobile, Alabama
  - Phoenix Childrens Hosp, Phoenix, Arizona
  - UCSD Med Ctr / Pediatrics / Clinical Sciences, La Jolla, California
  - Long Beach Memorial (Pediatric), Long Beach, California
  - Los Angeles County - USC Med Ctr, Los Angeles, California
  - Cedars Sinai / UCLA Med Ctr, Los Angeles, California
  - UCLA Med Ctr / Pediatric, Los Angeles, California
  - Harbor - UCLA Med Ctr / UCLA School of Medicine, Los Angeles, California
  - Children's Hosp of Denver, Denver, Colorado
  - Connecticut Children's Med Ctr, Farmington, Connecticut
  - Yale Univ Med School, New Haven, Connecticut
  - Howard Univ Hosp, Washington D.C., District of Columbia
  - North Broward Hosp District, Fort Lauderdale, Florida
  - Univ of Florida Gainesville, Gainesville, Florida
  - Univ of Florida Health Science Ctr / Pediatrics, Jacksonville, Florida
  - Univ of Miami / Jackson Memorial Hosp, Miami, Florida
  - Univ of Miami (Pediatric), Miami, Florida
  - Arnold Palmer Hosp for Children & Women, Orlando, Florida
  - Sacred Heart Children's Hosp / CMS of Florida, Pensacola, Florida
  - Palm Beach County Health Dept, Riviera Beach, Florida
  - Univ of South Florida, Tampa, Florida
  - Emory Univ Hosp / Pediatrics, Atlanta, Georgia
  - Med College of Georgia, Augusta, Georgia
  - The Med Ctr Inc, Columbus, Georgia
  - Univ of Illinois College of Medicine / Pediatrics, Chicago, Illinois
  - Chicago Children's Memorial Hosp, Chicago, Illinois
  - Tulane Univ / Charity Hosp of New Orleans, New Orleans, Louisiana
  - Univ of Maryland at Baltimore / Univ Med Ctr, Baltimore, Maryland
  - Johns Hopkins Hosp - Pediatric, Baltimore, Maryland
  - Children's Hosp of Boston, Boston, Massachusetts
  - Baystate Med Ctr of Springfield, Springfield, Massachusetts
  - Children's Hosp of Michigan, Detroit, Michigan
  - Univ of Mississippi Med Ctr, Jackson, Mississippi
  - Washington Univ School of Medicine, St Louis, Missouri
  - Cooper Hosp - Univ Med Ctr / UMDNJ - New Jersey Med Schl, Camden, New Jersey
  - UMDNJ - Robert Wood Johnson Med School / Pediatrics, New Brunswick, New Jersey
  - St Peter's Med Ctr, New Brunswick, New Jersey
  - Univ of Medicine & Dentistry of New Jersey / Univ Hosp, Newark, New Jersey
  - Saint Joseph's Hosp and Med Ctr/UMDNJ - New Jersey Med Schl, Newark, New Jersey
  - Children's Hosp at Albany Med Ctr, Albany, New York
  - SUNY - Brooklyn, Brooklyn, New York
  - North Shore Univ Hosp, Great Neck, New York
  - Bellevue Hosp / New York Univ Med Ctr, New York, New York
  - Cornell Univ Med College, New York, New York
  - Metropolitan Hosp Ctr, New York, New York
  - Columbia Presbyterian Med Ctr, New York, New York
  - Harlem Hosp Ctr, New York, New York
  - Univ of Rochester Med Ctr, Rochester, New York
  - State Univ of New York at Stony Brook, Stony Brook, New York
  - SUNY Health Sciences Ctr at Syracuse / Pediatrics, Syracuse, New York
  - Bronx Lebanon Hosp Ctr, The Bronx, New York
  - Duke Univ Med Ctr, Durham, North Carolina
  - Univ of North Carolina at Chapel Hill / Duke Univ Med Ctr, Durham, North Carolina
  - Columbus Children's Hosp, Columbus, Ohio
  - Med Univ of South Carolina, Charleston, South Carolina
  - Univ of South Carolina School of Med, Columbia, South Carolina
  - Children's Med Ctr of Dallas, Dallas, Texas
  - Texas Children's Hosp / Baylor Univ, Houston, Texas
  - Univ of Texas Health Sciences Ctr, San Antonio, Texas
  - Med College of Virginia, Richmond, Virginia
  - Children's Hospital & Medical Center / Seattle ACTU, Seattle, Washington
- Brazil (3):
  - Federal University of Minas, Dept. of Pediatrics, Belo Horizonte-MG
  - Hosp dos Servidores do Estado, Rio de Janeiro
  - Hosp Univ Clementino Fraga Filho, Rio de Janeiro RJ
- Puerto Rico (6):
  - Ramon Ruiz Arnau Univ Hosp / Pediatrics, Bayamón
  - Caguas Regional Hosp, Caguas
  - Mayguez Med Ctr / Regional Immunology Clinic, Mayguez
  - Ponce Univ Hosp, Ponce
  - Univ of Puerto Rico / Univ Children's Hosp AIDS, San Juan
  - San Juan City Hosp, San Juan
- Princess Margaret Hosp, Nassau, The Bahamas

REFERENCES:
- [Background] Kaiser M, Hagopian J, Ernestine J, Moye J, Fowler M, Nesel C. Providing access to HIV-research opportunities for disenfranchised populations. Int Conf AIDS. 1998;12:845-6 (abstract no 42358)